CLINICAL TRIAL: NCT00527917
Title: A Multi-Center, Randomized, Double-Blind, Parallel Group Evaluation of the Efficacy and Safety of Uracyst® (Intravesical Sodium Chondroitin Sulfate) Versus Vehicle Placebo in Patients With Interstitial Cystitis/Painful Bladder Syndrome.
Brief Title: A Pilot Clinical Investigation of the Efficacy and Safety of Uracyst® Versus Placebo in Patients With Interstitial Cystitis/Painful Bladder Syndrome.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Watson Pharmaceuticals (Industry)
Responsible Party: Gary Hoel Ph.D. Executive Director, Watson Laboratories Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UR07001
Record Dates: First submitted 2007-09-07; First posted 2007-09-11 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2009-12

CONDITIONS: Interstitial Cystitis
Keywords: IC/PBS; Interstitial Cystitis/Painful Bladder Syndrome
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Equipment and Supplies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Uracyst (Experimental): Sodium chondroitin sulfate
  Interventions: Device: Uracyst
- Placebo (Placebo Comparator): placebo
  Interventions: Device: placebo

INTERVENTIONS:
Device: placebo — bladder instillation
  Other Names: device vehicle
  Arms: Placebo
Device: Uracyst — 20 ml sterile solution for weekly intravesical instillation
  Other Names: sodium chondroitin sulfate
  Arms: Uracyst

SUMMARY:
This is a pilot clinical investigation. Patients who meet the eligibility criteria and provide signed informed consent will be randomized to receive either an active product (Uracyst®) or placebo intravesically via a bladder catheter weekly for 6 weeks, followed by 6 weeks of follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Are female of male patient 18 years or older
* Have been previously diagnosed with IC/PBS.
* Are willing to provide informed consent
* Available for the duration of the study including treatment and follow-up (12 weeks)

Exclusion Criteria:

* Pregnant or lactating female.
* Are currently or have previously received investigational drugs within thirty (30) days of screening.
* Previous therapy for IC/PBS
* Have any medical condition/disease that could interfere with patient compliance or interfere with interpretation of the study results.
* Are unable or unwilling to comply with protocol requirements
* Are unable to read, understand, and provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2007-09; Primary Completion 2008-06 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline to 6 weeks in Global Response Assessment instrument (GRA)score. The GRA evaluates symptoms of intersticial cystitis | Baseline to 6 weeks

SECONDARY OUTCOMES:
Adverse event assessments | Throughout the study, first instillation to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Keshava Kumar, PhD, Study Director — Watson Pharmaceuticals
Locations (13):
- Canada (13):
  - Surrey, British Columbia
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Kentville, Nova Scotia
  - Barrie, Ontario
  - Brantford, Ontario
  - Guelph, Ontario
  - Kingston, Ontario
  - Kitchener, Ontario
  - Newmarket, Ontario
  - North Bay, Ontario
  - Thunder Bay, Ontario
  - Toronto, Ontario